CLINICAL TRIAL: NCT00890786
Title: A Pilot Study of Bevacizumab-Based Therapy in Patients With Newly Diagnosed High-Grade Gliomas and Diffuse Intrinsic Pontine Gliomas
Brief Title: A Study of Bevacizumab Therapy in Patients With Newly Diagnosed High-Grade Gliomas and Diffuse Intrinsic Pontine Gliomas
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGG
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Newly Diagnosed High-Grade Gliomas; Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — Temozolomide; Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HGG (Experimental): Temozolomide, Bevacizumab, and Irinotecan according to the treatment schedule in the intervention section.
  Interventions: Drug: Temozolomide; Drug: Bevacizumab; Drug: Irinotecan
- DIPG (Experimental): Temozolomide, Bevacizumab, and Irinotecan according to the treatment schedule in the interventions section.
  Interventions: Drug: Temozolomide; Drug: Bevacizumab; Drug: Irinotecan

INTERVENTIONS:
Drug: Temozolomide — High Grade Glioma Temozolomide during radiotherapy: 90mg/m2/day PO daily (for patients ≤ 18 years of age); 75mg/m2/day PO daily (for patients ≥ 19 years of age); must begin by Day 5 of radiotherapy for a total of 42 days consecutively.
  High Grade Glioma Temozolomide during maintenance chemotherapy: 150mg/m2/day PO on Days 1-5.
  Other Names: Temodar
Drug: Bevacizumab — High Grade Glioma Bevacizumab during radiotherapy: 10 mg/kg as a 90 minute infusion on Day 22 (± 2 days)and Day 36 (± 2 days) of radiotherapy.
  High Grade Glioma Bevacizumab during maintenance chemotherapy:10 mg/kg as a 90 minute infusion on Day 1 (+ 2 days)and Day 15 (± 2 days) of each course.
  Diffuse Intrinsic Pontine Gliomas Bevacizumab during radiotherapy: 10 mg/kg as a 90 minute infusion on Days 1 (+ 2 days),15, 29, and 43(±2 days for all 3 doses) of radiotherapy.
  Diffuse Intrinsic Pontine Gliomas Bevacizumab during maintenance chemotherapy: 10 mg/kg as a 90 minute infusion on Day 1 (+2 days)and 15 (±2 days).
  Other Names: Avastin
Drug: Irinotecan — High Grade Glioma Irinotecan during maintenance chemotherapy:125 mg/m2/day IV over 90 minutes on Days 1 (+ 2 days)and 15 (±2 days) of each course, given no sooner than one hour after temozolomide on Day 1.
  Diffuse Intrinsic Pontine Gliomas Irinotecan maintenance chemotherapy: 125 mg/m2/day IV on Day 1 (+2 days)and Day 15 (±2 days).
  Other Names: Camptosar

SUMMARY:
The outcome for children with high-grade gliomas and diffuse intrinsic brainstem gliomas remains poor despite the use of multi-modal therapy with surgery, radiation therapy and chemotherapy.

DETAILED DESCRIPTION:
Novel therapies are needed to improve the outcome of these children. Recent studies have demonstrated very promising results of treatment with bevacizumab/irinotecan in patients with recurrent high grade gliomas. Based on these promising results, and the tolerability of the irinotecan and bevacizumab in children with recurrent CNS malignancies both anecdotally and in a study conducted by the Pediatric Brain Tumor Consortium, we have designed a novel study incorporating concurrent radiation therapy with bevacizumab ± temozolomide followed by bevacizumab, irinotecan ±temozolomide in patients with newly diagnosed high-grade gliomas and diffuse intrinsic pontine gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 3 years of age and ≤ 30 years of age at the time of study entry.
* Diagnosis:

  * High-grade glioma;Patients must have had histologically verified anaplastic astrocytoma, glioblastoma multiforme or gliosarcoma.Patients with primary spinal cord tumors are eligible.
  * Diffuse intrinsic pontine glioma (DIPG) are eligible.
* Performance Level: Karnofsky ≥ 50% for patients > 10 years of age and Lansky ≥ 50 for patients ≤ 10 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Prior Therapy: no prior anticancer therapy.
* Concomitant Medications: The use of steroids is permissible.
* Organ Function Requirements All patients must have adequate organ function as defined below.

  * Adequate Bone Marrow Function
  * Adequate Renal Function
  * Adequate Liver Function
* Adequate Blood Clotting Defined As: INR, Fibrinogen, and PTT < Grade 2
* Central nervous system function. Patients with seizures may be enrolled if the seizures are well-controlled with non-enzyme inducing anticonvulsants.
* Informed Consent. Patients and/or parents/legal guardians must have signed an informed consent.

Exclusion Criteria:

* Patients with metastatic disease (i.e. M+ disease, or disease anywhere other than primary site).
* Patients with evidence of a new intracranial hemorrhage that is larger than a punctate size on baseline MRI scan.
* Allergies: Patients with a history of allergic reaction to Chinese hamster ovary cell products, or other recombinant human antibodies.
* Pregnant or breast feeding women will not be entered on this study.
* Patients of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study.
* Infection: Patients who require IV antibiotics at time of enrollment, or who are currently receiving treatment for Clostridium difficile infection are excluded.
* Thrombosis: Patients must not have been previously diagnosed with a deep venous or arterial thrombosis (including pulmonary embolism), and must not have a known thrombophilic condition.
* Serious or Non-Healing Wounds
* Surgical Procedures: Patients who have had major surgery should not receive the first dose of bevacizumab until 28 days after major surgery.
* Patients with uncontrolled systemic hypertension.
* Proteinuria with a urine protein (albumin)/creatinine ratio of ≥1.0.

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2009-05; Primary Completion 2014-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To determine the toxicities and feasibility of the proposed treatment regimen in patients with high-grade glioma and diffuse intrinsic brainstem glioma | 2-3 years

SECONDARY OUTCOMES:
To determine 1-year EFS, median PFS and median OS in newly diagnosed patients with high-grade glioma treated with radiotherapy and concurrent temozolomide, bevacizumab followed by bevacizumab, irinotecan and temozolomide for 12 courses | 2-3 years
To determine the 1-year EFS, median PFS and median OS in newly diagnosed patients with diffuse intrinsic brainstem glioma treated with radiotherapy and concurrent bevacizumab followed by bevacizumab and irinotecan for 12 courses | 2-3 years
To estimate blood levels of VEGF in circulating endothelial cells in patients at different time points | 2-3 years
To document changes in MR perfusion and diffusion within 24-48 hours after the 2nd dose of bevacizumab during radiotherapy | 2-3 years
To correlate functional changes in tumor with responses to treatment using MR diffusion/perfusion imaging | 2-3 years
To correlate the results of the biology studies in serum or tumor with PFS | 2-3 years
To conduct gene expression profiling, CGH and SNP arrays in patients with high-grade gliomas | 2-3 years
To assess telomerase activity, hTert expression, and telomere length in patients with high-grade gliomas | 2-3 years
To assess the health-related quality of life of patients by parent report, and when possible, patient report at key points in therapy | 2-3 years
To assess functional abilities and level of independence of patients during and following treatment | 2-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Fouladi, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No